CLINICAL TRIAL: NCT01861873
Title: Phase 2 Study: Functional Treatment Planning Utilizing 18-FDGal PET/CT in SBRT for Liver Metastases
Brief Title: Functional Treatment Planning Utilizing 18-FDGal PET/CT in SBRT for Liver Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210982
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Liver Metastases
Keywords: liver function; galactose; 18-F-deoxy-galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- liver metastases (Other): measuring liver function by PET/CT at patients where SBRT is planned for liver metastases
  Interventions: Other: measuring liver function by 18-FDGal PET/CT

INTERVENTIONS:
Other: measuring liver function by 18-FDGal PET/CT

SUMMARY:
Background: Anatomical (traditional) stereotactic body radio therapy(SBRT) treatment planning assumes homogenous distribution of function in the normal liver tissue. In functional treatment planning, additional information on distribution of the function derived from functional imaging of normal tissue is taken into account. by functional treatment planning it becomes possible to prioritize and spare the best functioning part of an organ.

Aim: To test whether functional treatment planning based on 18-FDGal PET/CT may spare the best functioning liver tissue.

Endpoints: Reduction in hepatic systemic clearance (K) in the dynamic 18-FDGal PET/CT scan one month after SBRT compared to the baseline status in sub-volumes recieving 15 Gy or higher. Secondly, the investigators will evaluate the toxicity to SBRT by a toxicity scoring system that includes biochemical measures as well as symptomatic scores.

ELIGIBILITY:
Inclusion Criteria:

* Performance status >2
* liver metastases refereed for SBRT

Exclusion Criteria:

* pregnancy
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
volumetric uptake values of 18-FDGal will be measured and the 18-FDGal PET/CT one month after stereotactic body radioation therapy will be compared to the baseline status in sub-volumes receiving more than 15 Gy | up to 2 years

SECONDARY OUTCOMES:
evaluate toxicity to SBRT by toxicity scoring system that includes biochemical measures as well as symptomatic scores. | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark